CLINICAL TRIAL: NCT05547750
Title: Effect of Vitamin K2 in the Treatment of Nocturnal Leg Cramps in Older Population: Study Protocol of a Randomized, Double-blind, Controlled Trial
Brief Title: Effect of Vitamin K2 in the Treatment of Nocturnal Leg Cramps in Older Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Collaborators: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, Ying Li, Chief of hematology department, The Third People's Hospital of Chengdu
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-S17
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Nocturnal Leg Cramps
Keywords: Nocturnal Leg Cramps; Vitamin K2; older population
MeSH Terms: conditions — Sleep-Wake Transition Disorders | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be classified into two intervention groups at a ratio of 1:1, using a computer-generated randomized sequence with varying unknown block sizes for all study centers without stratification. A research assistant not involved in clinical care and participant evaluations will prepare sequentially numbered, opaque, sealed envelopes based on a random list and ensure that anyone will not access or influence the allocation data. The participants, outcome assessor, and statistician will be blinded to group allocation and not involved in the treatment procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin K2 arm (Experimental): The vitamin K2 arm takes vitamin K2 180 μg/day at bedtime for 8 weeks.
  Interventions: Drug: Vitamin K2
- Placebo (Placebo Comparator): The placebo group takes a placebo at bedtime for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin K2 — Vitamin K2 is a fat-soluble and one of the body's indispensable vitamins. It is mainly synthesized by gut bacteria in the body and plays a role in the mitochondrial electron transport chain. It boosts calcium metabolism, acts on osteoblasts, and promotes bone tissue calcification. It also inhibits osteoclasts from causing bone resorption, thus increasing bone density, and preventing osteoporosis. Furthermore, it regulates the use of calcium and promotes the inhibition of vascular calcification by matrix Gla protein (MGP) activity. Vitamin K2 supplementation at recommended dosage does not affect vitamin K-dependent coagulation factors' activity. It does not enhance the carboxylation of prothrombin in healthy individuals. Vitamin K2 administration does not alter the hemostatic balance in healthy populations without anticoagulation treatment. Thus, vitamin K2 is deemed to have a good safety profile.
  Arms: vitamin K2 arm
Drug: Placebo — Similar-looking placebo tablets
  Arms: Placebo

SUMMARY:
Nocturnal leg cramps (NLCs) are sudden contractions of the leg muscles, usually in the posterior calf muscles at night, affecting sleep quality. Because the precise pathophysiology of NCLs is unclear, different interventions have been proposed. There is conflicting evidence regarding the efficacy of conventional interventions in preventing cramps. Thus, the present study aims to investigate the effects of vitamin K2 for NLCs in a prospective randomized, double-blind, controlled trial.

DETAILED DESCRIPTION:
Nocturnal leg cramps (NLCs) are spontaneous contractions of muscles. The gastrocnemius is commonly involved, lasting from a few seconds to a few minutes. Patients might wake up with pain during attacks, making it difficult to sleep for a short period. It commonly occurs >60-year-old. The medical history and physical examination are usually sufficient to differentiate nocturnal leg cramps from other conditions, such as restless legs syndrome, claudication, myositis, and peripheral neuropathy. Factors that may lead to leg cramps attacks include hemodialysis, electrolyte imbalance, metabolic disorders, and congenital disorders. The cramps can be relieved by passive stretching of the gastrocnemius and deep tissue massage, but such prevention is limited, especially in patients with refractory muscle cramps. Quinine has been shown to be effective in treating NLCs but is not recommended by the US Food and Drug Administration due to severe side effects. Magnesium supplements are often used as a preventative treatment for NLCs; however, their effectiveness is controversial. Magnesium supplements are widely marketed for the prophylaxis of NLCs since a double-blind, placebo-controlled study proved their effectiveness in pregnant women. However, magnesium administration did not show significant benefits in NLCs in double-blind, placebo-controlled studies. Meta-analysis of some randomized control trials (RCTs) showed that magnesium therapy did not appear to be effective in the treatment of NLCs in the general population, but may have a negligible effect in pregnant women. Therefore, seeking new approaches to manage NLCs is imperative.

Vitamin K is a fat-soluble vitamin involved in carboxylation and activating several dependent proteins. It is found in two isoforms (phylloquinone (vitamin K1) and menaquinone (vitamin K2)) that differ in length and degree of saturation of the side chain. In addition to their role in coagulation, vitamin K-dependent proteins are involved in vascular calcification and osteoporosis physiology. Accumulating evidence has shown the beneficial effects of vitamin K2 supplementation on cardiovascular and bone health.

Another study revealed that vitamin K3 relieved muscle cramps by effectuating the voltage-dependent calcium channels to release the calcium stored in the cells, thus reducing the frequency of muscular contractions. To the best of our knowledge, no study has yet investigated the efficacy of vitamin K in NLCs. In addition, vitamin K2 has a good safety profile compared to other medications. Our pilot study demonstrated that vitamin K2 supplementation decreases the frequency, duration, and severity of muscle cramps in hemodialysis patients. To further investigate the efficacy and safety of vitamin K2 in NLCs, we designed this prospective, multicenter, randomized, double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

1. Unexplained cramps occurred two or more times in 2 weeks.
2. Age ≥65-year-old.

Exclusion criteria

1. Cramps caused by specific metabolic diseases and specific neuropathies (hypothyroidism, hemodialysis, hypoglycemia, alcoholism, amyotrophic lateral sclerosis, and poliomyelitis complications, lumbar spinal stenosis, Parkinson's disease, radiculopathies, and motor neuron diseases);
2. Suffering from malignant tumors (breast cancer, prostate cancer, lymphoma, and multiple myeloma);
3. Taking diuretics, or vitamin K antagonist;
4. Taking supplements with vitamin K2 within 2 months before enrollment;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The number of NLCs attacks | Comparing frequency differences between vitamin K2 and placebo treatment phases of NLCs in a 8 weeks investigation
  The mean number of NLC attacks per week

SECONDARY OUTCOMES:
The duration of NLCs | During the 8 weeks of investigation, the differences in the duration during NLCs attacks will record in the trial compared to vitamin K2- and placebo-treated arms
  Duration of muscle cramps in minutes
The severity of NLCs | During the 8 weeks of investigation, pain severity during NLCs attacks is recorded in the trial and compared to vitamin K2- and placebo-treated arms
  The severity of muscle cramps using a 1-10 analog scale（1-3 points, mild pain, tolerable, does not affect sleep; 4-6 points, moderate pain, affects sleep, also tolerable; 7-10 points, sharp pain, intolerable.）

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Third People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan J, Zhu R, Li Y, Wang L, Liao S, Cheng L, Mao L, Jing D. Vitamin K2 in Managing Nocturnal Leg Cramps: A Randomized Clinical Trial. JAMA Intern Med. 2024 Dec 1;184(12):1443-1447. doi: 10.1001/jamainternmed.2024.5726. PMID 39466236
- [Derived] Li Y, Zhu R, Wang L, Tan J. Effect of vitamin K2 in the treatment of nocturnal leg cramps in the older population: Study protocol of a randomized, double-blind, controlled trial. Front Nutr. 2023 Feb 23;10:1119233. doi: 10.3389/fnut.2023.1119233. eCollection 2023. PMID 36908924